CLINICAL TRIAL: NCT02883621
Title: Comparison Between Standard Endoscopy and Cap Assisted Endoscopy for Diagnostic Yield in Esophagus
Brief Title: The Diagnostic Yield of Cap Assisted Upper Endoscopy in Esophagus
Acronym: Kappa-III
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Technical University of Munich (Other)
Collaborators: Klinikum Freising (Unknown); Klinikum Landshut-Achdorf (Unknown); Städtisches Klinikum Neuperlach (Unknown); Rotkreuzklinikum München gGmbH (Other); Gemeinschaftspraxis Dr. Schatke & Dr. Ott (Unknown); Gastroenterologische Fachpraxis Abdomen Prof. Dr. Manfred Kurjak (Unknown)
Responsible Party: Principal Investigator, Mohamed Abdelhafez, MD, Technical University of Munich
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 218/16 s
Record Dates: First submitted 2016-08-21; First posted 2016-08-30 (Estimated); Last update posted 2017-05-23 (Actual); Status verified 2017-05

CONDITIONS: Endoscopic Diagnosis in Esophagus
Keywords: upper endoscopy; cap assisted endoscopy; esophagus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group A (Active Comparator): subjects receive standard upper endoscopy
  Interventions: Procedure: standard upper endoscopy
- Group B (Experimental): subjects receive cap assisted upper endoscopy
  Interventions: Procedure: cap assisted upper endoscopy

INTERVENTIONS:
Procedure: cap assisted upper endoscopy — A soft plastic cap is attached to the tip of the scope to allow pressing of the folds and thus enhance the visualization.
  Other Names: cap fitted upper endoscopy
  Arms: Group B
Procedure: standard upper endoscopy — standard examination without using a cap
  Arms: Group A

SUMMARY:
Cap assisted colonoscopy, a simple technique of fixing a transparent plastic cap to the tip of the colonoscope, was proven to increase the adenoma detection rate during screening colonoscopy by helping to depress and flatten colonic folds, thereby improving visualization and decreasing blind mucosal areas. The usefulness of cap assisted upper endoscopy (CAE) is still under investigations. The aim of this study is to compare the diagnostic yield of the CAE to the standard endoscopy in esophagus.

ELIGIBILITY:
Inclusion Criteria:

* indication for upper endoscopy
* age over 18 years
* ability to provide informed consent

Exclusion Criteria:

* known or suspected upper gastrointestinal strictures
* upper gastrointestinal bleeding
* previous upper endoscopy during the last three months
* American Society of Anesthesiologists class III or higher

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1000 (Actual)
Dates: Start 2016-09; Primary Completion 2017-04 (Actual); Study Completion 2017-05-22 (Actual)

PRIMARY OUTCOMES:
Diagnostic yield in esophagus | 15 Minutes
  All endoscopic abnormalities in esophagus which are detected during the examination in both groups will be documented, analyzed and compared

SECONDARY OUTCOMES:
Overall diagnostic yield in upper gastrointestinal tract. | 15 Minutes
  All other endoscopic abnormalities outside the esophagus (stomach and duodenum) which are detected during the examination in both groups will be documented, analyzed and compared

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Abdelhafez, MD, Principal Investigator — II Medizinische Klinik am Klinikum rechts der Isar der Technischen Universität München
Locations (1):
- II Medizinische Klinik am Klinikum rechts der Isar der Technischen Universität München, Munich, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: No